CLINICAL TRIAL: NCT05935748
Title: A Phase 2 Trial to Evaluate the Safety and Efficacy of NKT2152 in Combination With Palbociclib (Doublet) and With Palbociclib and Sasanlimab (Triplet) in Subjects With Advanced or Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: Ph2 Study NKT2152 With Palbociclib & Sasanlimab in Subjects With Advanced Clear Cell Renal Cell Carcinoma (ccRcc)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated as a result of Sponsor portfolio reprioritization.
Sponsor: NiKang Therapeutics, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKT2152-202
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: ccRCC; Clear Cell Renal Cell Carcinoma; Kidney Cancer; Kidney Neoplasms; Renal Cancer; Renal Neoplasms; Recurrent Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Refractory Renal Cell Carcinoma; Advanced Renal Cell Carcinoma; Carcinoma; Neoplasms; Carcinoma, Renal Cell; Neoplasms, Glandular and Epithelial; Neoplasm by Histology; Adenocarcinoma; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Kidney Diseases; Urologic Diseases
Keywords: HIF2a; Hypoxia-inducible factor 2alpha; CDK4 inhibitor; CDK6 inhibitor; PD-1; immune checkpoint inhibitors
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Carcinoma; Neoplasms; Neoplasms, Glandular and Epithelial; Adenocarcinoma; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Kidney Diseases; Urologic Diseases | interventions — palbociclib

STUDY DESIGN:
Intervention Model Description: Lead-in/Dose Escalation (doublet & triplet combination) and Dose Expansion (doublet & triplet combination)
Masking Description: Randomization during Expansion phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lead-in Doublet combination (Experimental): Lead-in Doublet assesses safety of oral dosing NKT2152 at increasing dosage levels in combination with palbociclib to determine a recommended dose for expansion (RDE).
  Interventions: Drug: NKT2152; Drug: palbociclib
- Lead-in Triplet combination (Experimental): Lead-in Triplet assesses the safety of two doses of NKT2152 identified in the Doublet arm (RDE and RDE-1) by orally dosing ccRCC patients with NKT2152 in combination with palbociclib and sasanlimab
  Interventions: Drug: NKT2152; Drug: palbociclib; Other: sasanlimab
- Expansion Doublet combination (Experimental): Subjects randomized to Arm 1 will receive the Doublet combination (NKT2152 in combination with palbociclib) to provide an assessment of anti-tumor activity and to determine the RP2D.
  Interventions: Drug: NKT2152; Drug: palbociclib
- Expansion Triplet combination (Experimental): Subjects randomized to Arm 2 will receive the Triplet therapy (NKT2152 in combination with palbociclib and sasanlimab) to provide an assessment of anti-tumor activity and to determine the RP2D.
  Interventions: Drug: NKT2152; Drug: palbociclib; Other: sasanlimab

INTERVENTIONS:
Drug: NKT2152 — Oral HIF2a inhibitor
Drug: palbociclib — a cyclin-dependent kinases (CDK) 4 and 6 inhibitor
  Other Names: IBRANCE®
Other: sasanlimab — an immunoglobulin G4 (IgG4) monoclonal antibody that blocks PD-1; a solution for injection for subcutaneous administration
  Arms: Expansion Triplet combination; Lead-in Triplet combination

SUMMARY:
The goal of the Lead-in phase of the study is to evaluate the safety, efficacy, pharmacokinetics (PK) and determine recommended dose for expansion (RDE) of NKT2152 in combination with palbociclib (Doublet) and with palbociclib and sasanlimab (Triplet) in subjects with advanced or metastatic clear cell renal cell carcinoma (ccRCC) who received prior therapy. The goal of the Expansion phase of the study is to evaluate the safety, efficacy, PK at the selected RDE and identify the RP2D for NKT2152 in combination with palbociclib (Doublet) and with palbociclib and sasanlimab (Triplet) in subjects with advanced or metastatic clear cell renal cell carcinoma (ccRCC) who received prior therapy.

DETAILED DESCRIPTION:
This is a Phase 2 open-label, multicenter, global study of NKT2152. This study is designed as two phases: a Lead-in phase and an Expansion phase. Patients must be 18 years or older, with advanced or metastatic clear cell renal cell carcinoma (ccRCC). Eligible patients must have progressed or relapsed after at least 1 prior anti-vascular endothelial growth factor (VEGF)/VEGF receptor (VEGFR) systemic therapy and 1 immune checkpoint inhibitor (ICI) for advanced or metastatic ccRCC alone or in combination.

The Lead-in phase is designed as a dose escalation phase to evaluate the safety, efficacy, pharmacokinetics (PK) and determine recommended dose for expansion (RDE) of NKT2152 in combination with palbociclib and sasanlimab in advanced or metastatic ccRCC patients who received prior therapy.

The subsequent Expansion phase will evaluate the safety, efficacy, PK at the selected RDE and identify the RP2D for NKT2152 in combination with palbociclib and sasanlimab in advanced or metastatic ccRCC patients who received prior therapy.

ELIGIBILITY:
Inclusion Criteria:

* Must have locally advanced or metastatic ccRCC and have progressed or relapsed after at least 1 prior anti-VEGF/VEGFR systemic therapy and 1 ICI.
* Measurable disease per the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
* KPS score of at least 70%
* Able to swallow oral medications.

Exclusion Criteria:

* Active CNS metastases and/or carcinomatous meningitis
* Has had any major cardiovascular event within 6 months or clinically significant cardiovascular disease
* Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 3 months before administration of study drug.
* Has known HIV
* History of hepatitis B or known active hepatitis C infection
* Has received prior treatment with NKT2152, other HIF2α inhibitors, other CDK 4/6 inhibitors, palbociclib, or sasanlimab
* Radiation therapy for bone metastasis within 2 weeks, or any other external radiation therapy within 4 weeks before administration of the first dose of study treatment
* Corrected QT interval calculated by Fridericia formula (QTcF) > 480 ms within 28 days prior to first dose
* Hypoxia or requires intermittent or chronic supplemental oxygen or any chronic lung condition which has required supplemental oxygen in the past
* Has a history of interstitial lung disease
* Has any active or recent history of a known or suspected autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicity (DLT) events during the DLT monitoring period (first 28 days of dosing) in the Lead-in Phase | 28 days
  DLTs graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5 .0.
Objective Response Rate (ORR) determined by the Investigator | 1 years
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  PFS defined as the time from the date the participant started study drug to the date the participant experiences an event of disease progression or death.
Duration of Response (DOR) | 1 years
  Duration of overall response is defined as the time from the date of first documented CR or PR, assessed by investigator and based on RECIST v. 1.1, to the documented date of progressive disease (PD) or death, whichever occurred first.
Time to Response (TTR) | 1 years
  TTR is defined as the time from first dose to the first documented CR or PR which is subsequently confirmed.
Overall Survival (OS) | 2 years
  OS defined as the time from the date the participant started study drug to death for any reason.
Clinical Benefit Rate (CBR) | 1 years
  CBR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) or a stable disease (SD) of 8 weeks or longer based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Number of Participants with Adverse Events | 2 years
  An adverse event (AE) is defined as any untoward medical occurrence in a patient and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related.
Maximum observed plasma concentration (Cmax) of NKT2152 | 1 years
  Maximum observed plasma concentration (Cmax) of NKT2152
Time to maximum observed plasma concentration of NKT2152 (Tmax) | 1 years
  Time to maximum observed plasma concentration of NKT2152 (Tmax)
Observed trough concentration of NKT2152 (Ctrough) | 1 years
  Observed trough concentration of NKT2152 (Ctrough)
Area under the plasma concentration time curve (AUC0-t) of NKT2152, and accumulation ratio (RAC) | 1 years
  Area under the plasma concentration time curve (AUC0-t) of NKT2152, and accumulation ratio (RAC)
Maximum observed plasma concentration (Cmax) of palbociclib | 1 years
  Maximum observed plasma concentration (Cmax) of palbociclib
Time to maximum observed plasma concentration of palbociclib (Tmax) | 1 years
  Time to maximum observed plasma concentration of palbociclib (Tmax)
Observed trough concentration of palbociclib (Ctrough) | 1 years
  Observed trough concentration of palbociclib (Ctrough)
Area under the plasma concentration time curve (AUC0-t) of palbociclib, and accumulation ratio (RAC) | 1 years
  Area under the plasma concentration time curve (AUC0-t) of palbociclib, and accumulation ratio (RAC)
Observed trough concentration of sasanlimab (Ctrough) | 1 years
  Observed trough concentration of sasanlimab (Ctrough)
Maximum observed plasma concentration (Cmax) of sasanlimab | 1 years
  Maximum observed plasma concentration (Cmax) of sasanlimab

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California San Diego, La Jolla, California
  - Northwestern University - Feinberg School of Medicine, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan-Rogel Cancer Center, Ann Arbor, Michigan
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No
IPD are not planned to be shared at this time